CLINICAL TRIAL: NCT02439255
Title: Interactive Omics: Black Raspberry Metabolites and the Oral Microbiome in Smokers
Brief Title: Effect of Black Raspberry Phytochemicals on Oral Microbiome in Current Smokers and Non-smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Purnima Kumar, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-14135; NCI-2014-02622 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Healthy Subject; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Phytochemicals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I Black raspberry(BRB) nectar (Experimental): Participants receive BRB nectar PO QD for 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Dietary Supplement: Phytochemical; Other: Screening Questionnaire Administration
- Arm II (placebo nectar) (Placebo Comparator): Participants receive placebo nectar PO QD for 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Screening Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Phytochemical — Given black raspberry (BRB) nectar per oral (PO)
  Other Names: Phytonutrients
  Arms: Arm I Black raspberry(BRB) nectar
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo nectar)
Other: Screening Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies the effects of black raspberry compounds (phytochemicals) on the bacteria in the mouth (oral microbiome) of current smokers and non-smokers. The oral microbiome protects the body from pathogenic bacteria. Smoking alters the oral microbiome and may increase the susceptibility to cancer by modulating normal host-bacteria interactions. Black raspberry phytochemicals may protect the oral microbiome of smokers and may lower their risk of developing oral cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effect of black raspberry phytochemicals on community dynamics within oral biofilms.

II. Examine the effect of oral bacterial communities on metabolism of black raspberry phytochemicals in current and never smokers.

III. Evaluate the efficacy of black raspberry phytochemicals and their metabolites in reversing the effect of smoking on oral host-microbial interactions.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive bioactivity of black raspberry phytochemical-rich delivery vehicle (BRB nectar) orally (PO) once daily (QD) for 12 weeks.

ARM II: Participants receive placebo nectar PO QD for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be periodontally healthy; this is defined as all sites with attachment levels =< 2 mm and probing depths =< 3 mm) and caries-free, as evidenced by a DMF (decayed, missing, filled teeth) Index of less than 5
* Subject must be either a current smoker or a never smoker; to define a smoker, we will utilize the Centers for Disease Control definitions; any individual who is currently smoking and has smoked more than 100 cigarettes in their lifetime will be identified as a current smoker; smoking status will be assessed by a questionnaire; since only current and never smokers are included, it is not necessary to measure cotinine levels; the number of cigarettes smoked per day and years of smoking will be used to calculate pack-years, which will be used as a measure of tobacco exposure; a never smoker is defined as a person who never smoked, or smoked less than 100 cigarettes in their lifetime, and who has not had a cigarette in over ten years
* Agree to consume a standardized vitamin/mineral supplement and avoid other nutrition, dietary or alternative medications/supplements for the duration of the study
* Agree to follow a controlled ellagitannin/low polyphenolic diet and to document consumption of polyphenolic foods each day of the study using our easy to document daily form

Exclusion Criteria:

* Have history of oral cancer or carcinoma in-situ
* Have had antibiotic therapy or professional cleaning within the previous 3 months
* Require antibiotic therapy prior to oral cleaning
* Have an active metabolic or digestive illness that impact phytochemical absorption and metabolism, including: diabetes, malabsorptive disorders (Crohn's disease, documented celiac disease, etc.), renal insufficiency (creatinine [Cr] > 1.4), hepatic insufficiency (nonalcoholic steatohepatitis [NASH], cirrhosis, active viral hepatitis), hyper- or hypothyroidism, or short bowel syndrome
* Are alcohol consumers (defined as an average consumption of greater than 1 drink/day over one week [wk] [one drink = 1 oz. liquor, 12 oz. beer])
* Are taking immunosuppressant medications, bisphosphonates or steroid medications
* Currently undergoing treatment for cancer with chemotherapy, hormone therapy, radiation, or biological therapy
* Have a known allergy or food intolerance to ingredients in study products (black raspberries or other berries)
* Are planning to conceive, or are currently pregnant or lactating
* Have had any active oral lesions in the past month or currently have any oral disease or obvious open sores in the oral cavity or surrounding the oral opening
* Are taking any medications that have known impact on immune responses (e.g. nonsteroidal anti-inflammatory drugs [NSAIDs] for chronic pain) or are actively being investigated for the prevention of tobacco related cancers will not be acceptable; a single 81 mg aspirin per day will be acceptable

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the microbial shift | Baseline to 12 weeks
  The analyses of the microbial shift data will use a two-factor (smoking and berry treatment) ANOVA model with interaction on the post-treatment minus baseline differences between appropriately transformed data. Phylogenetic distances and community similarity and diversity will be computed from the sequence data. The sensitivity of the phylogenetic analysis to the uncertain knowledge of the phylogenetic relationships will be examined using draws from the posterior distribution of trees in a Mr. Bayes analysis.
Change of metabolite profile in saliva, urine, and blood using high-performance liquid chromatography-mass spectrometry | Baseline to up to 12 weeks
  The analyses of the metabolite endpoint will use a two-factor (smoking and berry treatment) analysis of variance (ANOVA) model with interaction on the post-treatment minus baseline differences between appropriately transformed data. The number of transcripts as well as the level of each transcript (transformed values) will be used to compute a Bray-Curtis similarity Index between the community profile post-treatment and the baseline profile.

SECONDARY OUTCOMES:
Food frequency (FF) using the Viocare FF Questionnaire | Week 0
  PROC MIXED repeated measures models will be used.
Gene expression levels using next generation sequencing (NGS) | Up to 12 weeks
  The presence and abundance of mucosal messenger ribonucleic acid transcripts will be computed from the NGD sequence data. Variance stabilizing transformation will be applied to gene expression levels. The significance of differences between the two groups over time is then studied as changes in this contrast for smokers versus non-smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Kumar, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu